CLINICAL TRIAL: NCT06540781
Title: Investigation of Wet Cupping Therapy Effect on Cerebral Oxygenation Levels by NIRS
Brief Title: The Efficacy of Wet Cupping Therapy on Cerebral Oxygenation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Karabuk University (Other)
Responsible Party: Principal Investigator, SULEYMAN ERSOY, Head of Family Medicine Department, Karabuk University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: WCT-11
Record Dates: First submitted 2024-08-02; First posted 2024-08-06 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-03

CONDITIONS: Cerebral Hypoxia
Keywords: Cerebral oxygenation; Wet cupping therapy; NIRS
MeSH Terms: conditions — Hypoxia, Brain

STUDY DESIGN:
Intervention Model Description: Single arm pretest-posttest interventional study
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention Group (Experimental): The intervention group will receive one session of WCT. Before, during and after the WCT application cerebral oxygenation levels will be measured by NIRS device.
  Interventions: Procedure: wet cupping therapy

INTERVENTIONS:
Procedure: wet cupping therapy — The cupping (WCT) procedure consists of five phases:
  Primary suction: Using a manual suction pump, air was drawn from glass cups that were positioned on the chosen locations. The skin and subcutaneous tissue swelled as a result of the cups' five minutes of skin contact.
  Area disinfection: After disinfecting the cupped areas with povidone-iodine, they were wiped with sterile gauze.
  Scarification: Using a sterile number 11 surgical blade, superficial incisions measuring 20-30 gauge in length and 1-2 mm in depth were made on the skin.
  Bloodletting and secondary suction: Once again applied to the scarified areas, the previously removed cups created suction using the manual pump which was previously mentioned. In order to fill the cups, blood was drawn from the skin's and subcutaneous tissue's capillaries.
  Removing and dressing: After 10 minutes, the cups filled with blood were removed. The application areas were wiped with sterile gauze, and dressings were applied.

SUMMARY:
The aim of this clinical trial is to investigate the efficacy of wet cupping therapy (WCT) on cerebral oxygenation using the NIRS device. With the demonstration of the positive effect of the WCT on cerebral oxygenation, it was aimed to use it effectively in stroke rehabilitation.

In the outpatient clinic setting, firstly the sensor pads of the NIRS device will be attached to the arcus superciliaris (GB14) under the tuber frontalis on both sides. After the measurement is initiated, WCT will be applied to the planum occipitale (DU 20) and to the pars squamosa (GB6-8) of the temporal bone on the sides. Measurement will continue for 10 minutes during and after the WCT application. NIRS and oxygenation measurement data will be compared before, during, and after the WCT application.

DETAILED DESCRIPTION:
The importance of NIRS is that it can detect differences in tissue oxygen uptake that cannot be routinely identified by existing methods (24). The ability of near-infrared (NIR; near infrared; wavelength 650 - 1100nm) light to penetrate tissues and to be absorbed by some chromophores (such as haemoglobin, cytochrome oxidase, bilirubin, urobilin) has formed the basis of regional cerebral oxygen saturation (rScO2) measurement (15). NIRS is a technique in which the amount of absorption of NIR light by chromophore molecules [such as oxyhaemoglobin (O2Hb) and deoxyhaemoglobin (HHb), cytochrome-c oxidase (CCO), myoglobin] is measured while passing through tissues (16). rScO2 values less than 40% or changes greater than 25% from baseline values may be a harbinger of cerebral ischaemia (17). Cerebral oximetry has attracted attention because it is easy to use and uncomplicated. NIRS should be used as a trend monitor.

In the current study, it is aimed to investigate the efficacy of wet cupping therapy (WCT) on cerebral oxygenation using the NIRS device. Following the enrollment of the healthy individuals, they will all receive one session of WCT. During the WCT application, the cerebral oxygenation levels will be measured with an NIRS device.

In the outpatient clinic setting, the NIRS device's sensor pads will be attached to the arcus superciliaris (GB14) under the tuber frontalis on both sides. After the measurement is initiated, WCT will be applied to the planum occipitale (DU 20) and the pars squamosa (GB6-8) of the temporal bone on the sides. Measurement will continue for 10 minutes during and after the WCT application. The data obtained by NIRS will be compared before, during, and after the WCT application so that we will be able to find out any possible effects of WCT on cerebral oxygenation.

ELIGIBILITY:
Inclusion Criteria:

* Healthy individual
* Age 18-65 years
* Consent to participate

Exclusion Criteria:

* Having received cupping therapy in the past 3 months
* Contraindications for WCT (such as hemoglobin level below 9.5 g/dL, bleeding disorders, receiving antithrombotic or antiplatelet therapy, INR value above 1.5),
* Coexisting chronic conditions and using any medication

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Oxygen levels | Just before WCT application and 10 minutes after the application
  Cerebral oxygenation levels measured by NIRS device

CONTACTS AND LOCATIONS:
Overall Officials: Ali R Benli, Study Chair — Kayseri research hospital
Locations (1):
- Kayseri City Hospital, Kayseri, Turkey (Türkiye)